Effect of Telerehabilitation Versus Conventional Physiotherapy on Quality of Life, Pain, and Functional Outcomes in Patients Following Rotator Cuff Surgery

NCT Number: Not assigned

Document Date: 24.01.2025

You are invited to participate in a research study. Participation is completely voluntary. Before deciding whether to join, please carefully read the following information explaining the purpose of the study, use of your personal data, study procedures, potential benefits, and risks. If you choose to participate, you will be asked to sign this Informed Consent Form. You may withdraw at any time without penalty or loss of benefits, and your decision will not affect your medical care.

## STUDY PURPOSE:

The study aims to evaluate the effectiveness of telerehabilitation in individuals who have undergone rotator cuff surgery. The impact of interventions on physical recovery, pain levels, and overall quality of life will be analyzed. Thirty participants are planned to be included.

#### STUDY PROCEDURES:

Participants will undergo assessment by a physiotherapist for pain, joint range of motion, and muscle strength. Functional assessments will include the Disabilities of Arm, Shoulder, and Hand Questionnaire (DASH), quality of life will be measured with the Western Ontario Rotator Cuff Index (WORC), and pain will be evaluated using the Visual Analog Scale (VAS).

Participants will be assigned to one of two groups: the telerehabilitation group (experimental) will receive home-based rehabilitation supervised online by a physiotherapist, and the control group will receive conventional face-to-face physiotherapy. Both groups will perform the same exercise program three times per week, including stretching, strengthening, and therapy sessions. Assessments will be repeated after the 8-week intervention.

## POTENTIAL BENEFITS:

Participation will contribute data to the scientific literature regarding telerehabilitation after rotator cuff surgery.

#### POTENTIAL RISKS:

There are no known physical or psychological risks; guidance will be provided based on treatment progress. Any discomfort should be reported to the research team.

| P | Α | RT | [C] | PA | NT | R | ES | SPC | N | IS | IR | II | TI | ΓIES | ٠ |
|---|---|----|-----|----|----|---|----|-----|---|----|----|----|----|------|---|

Participants should attend scheduled sessions, perform exercises, and provide accurate health information. Completion of questionnaires and physical assessments is required.

## CONFIDENTIALITY:

All personal information will be kept confidential and anonymized in any publications. Only authorized personnel such as the ethics committee may access original records for scientific and ethical review purposes.

# QUESTIONS:

For any questions or concerns during or after the study, please contact the study investigator.

## STUDY DURATION:

Participants will be involved for 8 weeks.

## CONSENT:

I have read and understood the above information, my questions have been answered, and I voluntarily agree to participate. I understand I may withdraw at any time without penalty.

| Signature: | Date: |
|------------|-------|